CLINICAL TRIAL: NCT03598582
Title: Biological Predictive Factors of Response to Erythropoiesis Stimulating Agent (ESA) in Low Risk Myelodysplastic Syndromes (MDS) Patients
Brief Title: Biological Predictive Factors of Response to ESA in Low Risk MDS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association pour la recherche sur les Affections Malignes en Immunologie Sanguine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RETA
Record Dates: First submitted 2018-05-26; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndromes; erythropoiesis stimulating agents; factors of response
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — epoetin zeta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- epoetin zeta (Other): Patients received epoetin zeta (Retacrit®) 40000UI/week subcutaneously during 12 weeks.
  Interventions: Drug: Epoetin Zeta

INTERVENTIONS:
Drug: Epoetin Zeta — Patients received epoetin zeta (Retacrit®) 40000UI/week subcutaneously during 12 weeks.
  Response has been evaluated at 12 weeks according to IWG 2006 criteria. Patients with response continued on epoetin zeta. In non-responders, the patients have been excluded from the protocol.
  Other Names: Retacrit

SUMMARY:
In this trial, the investigators would like to understand why a small percentage of patients will be refractory to ESA (independently of International prognostic scoring system (IPSS) and % of blasts). In a retrospective study of the "Groupe Francophone des Myélodysplasies (GFM)" , the investigators showed that about 43% of patients are refractory or will relapse after initial response to ESA and it has been shown that these patients have a poorer survival. The investigators plan to give a 12-week treatment of Epoetin alfa or zeta in low risk MDS patients and measure different biological factors to predict response to ESA:

* evaluation by flow cytometry before and after treatment of the degree of dyserythropoiesis and dysgranulopoiesis which could explain the primary resistance or loss of response of a subset of patients,
* screening by molecular biology of predictive factors of response to ESA,
* Iron homeostasis will be measured via hepcidin, GDF-15 and ferritin levels.

DETAILED DESCRIPTION:
Lower risk MDS patients, with LOW and INT-1 IPSS score, with anemia Hb<10g/dl, requiring or not Red blood cel (RBC) transfusions, treated by erythropoiesis stimulating agent (ESA) according to national French recommendations ( epoetin zeta 40000 UI/week in lower risk MDS, <10% blasts, with Hb<10g/dl and sEPO<500UI/l, for 12 weeks).

BM aspirates are collected prospectively at T0 and at W12 of ESA treatment.

BM aspirates will be collected prospectively at inclusion in all 70 patients, after 12 weeks, in 70 patients.

Fresh bone marrow samples will be centralized at Cochin hospital for flow cytometry analysis of dyserythropoiesis and gene sequencing (Hematology laboratory, Cochin, Paris). "Ogata flow cytometry score" will be assessed locally in Mulhouse, Creteil, Tours, Grenoble or Cochin. Patients have been reevaluated at week 12 by flow cytometry "Ogata score".

Blood plasma will be been collected for analysis of GDF-15 and hepcidin, and sent to Cochin (Institut Cochin, Paris). Hepcidin level was measured by LC-MS/MS method in Louis Mourier Hospital.

Red score analysis was done in a centralized manner in Cochin, according to the methods described previously. Basically, it was evaluated on CD36, CD71 CV and Hb level according to the gender.

Genomic studies and Bioinformatic analysis Mutations in a selected panel of 39 genes will be screened in the 70 samples by a Next-Generation Sequencing (NGS) assay.

Sample size justification and Statistical analysis Sample size computation was based on the secondary endpoint which was the response rate. The investigators expected a response rate of 50-60%, therefore about 30 patients will be responders and 30 patients non responders. With 10%-15% of non evaluable biological data, n=70 patients should be included.

ELIGIBILITY:
Inclusion Criteria:

> 18y patients

* with MDS subtypes :

  * refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), refractory anemia with excess of blasts (RAEB) with <10 % blasts (according to FAB classification) CMML with white blood cell (WBC) <13.000/mm3
  * RA, RARS, RCMD, RAEB-1, CMML-1 with WBC <13.000/mm3 (according to OMS classification), 5q- syndrome
  * Low int-1 IPSS score
* With hemoglobin (Hb)<10 g/dL or red blood cell transfusion (RBC) transfusion dependent
* treated by ESA according to national French recommendations
* without renal insufficiency
* with ECOG PERFORMANCE STATUS <2

Exclusion Criteria:

* higher risk MDS (IPSS intermediate-2 or high)
* CMML with >10 % of BM blasts or WBC>13.000/mm3
* Non-controlled hypertension
* Cardio-vascular disease :uncontrolled, angina pectoris, cardiac insufficiency,
* Renal insufficiency : Creatinine clearance<40ml/min
* EPO level>500UI/l
* Systemic infection or inflammatory chronic disease
* Serum folates<2 ng/mL or vitamin B12 <200 pg/mL
* Other causes of anemia (eg hemolysis, hemorrhage, iron deficiency)
* Pregnancy (positive betaHCG) or nursing
* Women of childbearing age without effective contraception why?
* Hypersensitivity to Darbepoietin alfa or other ESA
* Patient unable to understand the protocol or to follow adequately
* History of epilepsy
* History of thrombosis
* Concomitant thalidomide or lenalidomide treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Determination of the Red score on the prediction of response to ESA | 5 years
  The flow cytometry (FCM) "Red score" described by Mathis et al, Leukemia 2013, ranges from 0 to 7 and includes CD36 and CD71 CV and Hb levels.
Determination of Ogata FCM score on the prediction of response to ESA | 5 years
  The "Ogata FCM score" described by Ogata et al, Haematologica 2009, ranges from 0 to 4 and includes parameters of dysgranulopoiesis and excess of CD34+ blasts
Determination of the number of molecular gene mutations on the prediction of response to ESA | 5 years
  Gene mutations numbers, assessed by next generation sequencing on a 39 gene panel
Determination of GDF-15 levels on the prediction of response to ESA | 5 years
  Mean and median values of GDF15 (pg/ml) levels
Determination of hepcidin levels on the prediction of response to ESA | 5 years
  Mean and median values of hepcidin (ng/ml)

SECONDARY OUTCOMES:
Response rate to ESA | 5 years
  Response rate will be evaluated by IWG 2006 criteria of erythroid response.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PARK, MD, PHD, Principal Investigator — CHU Grenoble Alpes